CLINICAL TRIAL: NCT00005476
Title: Sociodemographic Regulation of Cardiovascular Function and Structure
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 4960; R01HL056622 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-07-29 (Estimated); Status verified 2009-05

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Hypertension
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Hypertension

SUMMARY:
To establish the aspects of ethnicity that are associated with the differential expression of cardiovascular disease processes in African Americans and Caucasian Americans twin children.

DETAILED DESCRIPTION:
BACKGROUND:

Given increasing awareness of the extent to which environments typically faced by ethnic groups differ, environmental influence on these processes may be an important factor that is an aspect of ethnicity. Socioeconomic status (SES) is a useful index of such environments and is associated with cardiovascular disease (CVD). Since behavior is one pathway through which SES influences are thought to be expressed in disease, this study focuses specifically on stress responsivity, which is thought to be linked to the pathophysiology of CVD. Since such disease has its antecedents in childhood, a multiethnic pediatric sample is employed. In addition, the subject sample consists of twins. Investigation of the impact of environments on the expression of CVD can be achieved only with proper control for biological influences.

DESIGN NARRATIVE:

Subjects completed three laboratory stressors: a video game task, a structured social interview, and the cold pressor. Stress responsivity was assessed, with particular interest being paid to systemic vascular resistance (SVR). Left ventricular mass (LVM) was also assessed. Sophisticated environmentally and genetically informative analyses permitted quantification of environmental impact upon systemic vascular resistance responsivity and left ventricular mass. It was hypothesized that environmental influences (SES) accounted for a greater proportion of the variance in systemic vascular resistance responsivity and left ventricular mass in African Americans than Caucasian Americans. The hypothesis that systemic vascular resistance responsivity was a pathway through which SES exerted its influence on left ventricular mass was also tested.

The study has been extended through November 2005 to continue examination of the investigator's Twin CV Health cohort (519 pairs of twins who will be 14 to 25 years old). The study provides the unique opportunity to better understand the effects of sodium ion (Na+) retention as a mechanism augmenting systemic vascular resistance responsivity (SVR) and changes in vascular function (i.e., endothelium dependent arterial dilation; EDAD), ventricular structure (i.e., left ventricular mass; LVM) and 24-hour ambulatory BP (ABP). The specific aims are to determine: 1) To what extent is environmental stress related to stress induced Na+ retention, SVR responsivity and preclinical markers of essential hypertension risk and are these relationships stronger in African Americans than Caucasian Americans; 2) Whether stress induced Na+ retention is a pathway linking environmental stress with preclinical markers of essential hypertension risk; and 3) Whether behavioral factors (i.e. John Henryism, anger expression, social support, physical activity) moderate effects of environmental stress on stress induced Na+ retention and/or SVR responsivity and in the preclinical markers of essential hypertension risk, particularly in African Americans.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1996-09; Primary Completion 2005-11 (Actual); Study Completion 2005-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frank Treiber — Augusta University

REFERENCES:
- [Background] Jackson RW, Snieder H, Davis H, Treiber FA. Determination of twin zygosity: a comparison of DNA with various questionnaire indices. Twin Res. 2001 Feb;4(1):12-8. doi: 10.1375/1369052012092. PMID 11665319
- [Background] Davis CL, Kapuku G, Snieder H, Kumar M, Treiber FA. Insulin resistance syndrome and left ventricular mass in healthy young people. Am J Med Sci. 2002 Aug;324(2):72-5. doi: 10.1097/00000441-200208000-00005. PMID 12186110
- [Background] Snieder H, Harshfield GA, Barbeau P, Pollock DM, Pollock JS, Treiber FA. Dissecting the genetic architecture of the cardiovascular and renal stress response. Biol Psychol. 2002 Oct;61(1-2):73-95. doi: 10.1016/s0301-0511(02)00053-4. PMID 12385670
- [Background] Barbeau P, Litaker MS, Jackson RW, Treiber FA. A tyrosine hydroxylase microsatellite and hemodynamic response to stress in a multi-ethnic sample of youth. Ethn Dis. 2003 Spring;13(2):186-92. PMID 12785414
- [Background] Snieder H, Treiber FA. The Georgia Cardiovascular Twin Study. Twin Res. 2002 Oct;5(5):497-8. doi: 10.1375/136905202320906354. PMID 12537884
- [Background] Snieder H, Dong Y, Barbeau P, Harshfield GA, Dalageogou C, Zhu H, Carter ND, Treiber FA. Beta2-adrenergic receptor gene and resting hemodynamics in European and African American youth. Am J Hypertens. 2002 Nov;15(11):973-9. doi: 10.1016/s0895-7061(02)02991-6. PMID 12441217
- [Background] Snieder H, Harshfield GA, Treiber FA. Heritability of blood pressure and hemodynamics in African- and European-American youth. Hypertension. 2003 Jun;41(6):1196-201. doi: 10.1161/01.HYP.0000072269.19820.0D. Epub 2003 Apr 28. PMID 12719445
- [Background] Wang X, Trivedi R, Treiber F, Snieder H. Genetic and environmental influences on anger expression, John Henryism, and stressful life events: the Georgia Cardiovascular Twin Study. Psychosom Med. 2005 Jan-Feb;67(1):16-23. doi: 10.1097/01.psy.0000146331.10104.d4. PMID 15673619
- [Background] Iliadou A, Snieder H, Wang X, Treiber FA, Davis CL. Heritabilities of lipids in young European American and African American twins. Twin Res Hum Genet. 2005 Oct;8(5):492-8. doi: 10.1375/183242705774310187. PMID 16212838
- [Background] Imumorin IG, Dong Y, Zhu H, Poole JC, Harshfield GA, Treiber FA, Snieder H. A gene-environment interaction model of stress-induced hypertension. Cardiovasc Toxicol. 2005;5(2):109-32. doi: 10.1385/ct:5:2:109. PMID 16046788